CLINICAL TRIAL: NCT00673959
Title: Acute Comfort of Lubricant Eye Drop FID 111421
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-08
Record Dates: First submitted 2008-05-02; First posted 2008-05-07 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubricant Eye Drop FID 111421 (Experimental): Lubricant Eye Drop FID 111421 1 drop each eye one time
  Interventions: Other: Lubricant Eye Drop FID 111421
- Optive Lubricant Eye Drop (Active Comparator): Optive Lubricant Eye Drop 1 drop each eye one time
  Interventions: Other: Optive Lubricant Eye Drop

INTERVENTIONS:
Other: Lubricant Eye Drop FID 111421 — Lubricant Eye Drop FID 111421 1 drop each eye one time
  Arms: Lubricant Eye Drop FID 111421
Other: Optive Lubricant Eye Drop — Optive Lubricant Eye Drop 1 drop each eye one time
  Arms: Optive Lubricant Eye Drop

SUMMARY:
To evaluate the acute comfort and blurring profile between two artificial tears products in dry eye patients

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye
* Must not have worn contact lenses for 1 week preceding enrollment

Exclusion Criteria:

* Age related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 Dry Eye Subjects
Pre-assignment Details: Randomized, double-masked, crossover
Groups:
- Lubricant Drops, Then Optive Drops: Patients received Lubricant Drops first, then received Optive Drops
- Optive Drops, Then Lubricant Drops: Patients received Optive Drops first, then received Lubricant Drops
Period: Overall Study
Arm/Group | Lubricant Drops, Then Optive Drops | Optive Drops, Then Lubricant Drops
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Drop Comfort Upon Instillation
Description: Drop comfort grading scale is a scale from 0 to 9, with 0 meaning most comfortable and 9 meaning most uncomfortable.
Time Frame: upon instillation
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lubricant Eye Drop FID 111421 | Optive Lubricant Eye Drop
Number analyzed (Participants) | 20 | 20
Units on a scale | 1.7 (1.8) | 1.3 (1.4)

ADVERSE EVENTS:
Arm/Group | Lubricant Eye Drop FID 111421 | Optive Lubricant Eye Drop
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI should hold confidential, and not disclose directly or indirectly to any third party onther than Contractors, the data arising out of the study.